CLINICAL TRIAL: NCT05438108
Title: An Open, Single-arm, Exploratory Study of SBRT Sequential CapeOX Chemotherapy Combined With Bevacizumab and Sintilimab in First-line Treatment of Metastatic Colorectal Cancer
Brief Title: SBRT Sequential CapeOX Regimen Combined With Bevacizumab and Sintilimab in First-line Treatment of mCRC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianglin Yuan, professor, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJCC013
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Metastatic Colorectal Cancer
Keywords: mCRC; SBRT; chemotherapy; immune checkpoint inhibitor
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; sintilimab

STUDY DESIGN:
Intervention Model Description: SBRT Sequential CapeOX Regimen Combined With Bevacizumab and Sintilimab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT sequential chemotherapy, bevacizumab and sitilimab (Experimental)
  Interventions: Combination Product: SBRT Sequential CapeOX Regimen Combined With Bevacizumab and Sintilimab

INTERVENTIONS:
Combination Product: SBRT Sequential CapeOX Regimen Combined With Bevacizumab and Sintilimab — SBRT Sequential CapeOX Regimen Chemotherapy Combined With Bevacizumab and Sintilimab

SUMMARY:
Immune checkpoint inhibitors have a poor effect on MSS colorectal cancer. Studies have shown that SBRT, chemotherapy and anti-vascular therapy can enhance the anti-tumor effect of PD-1 antibody. This is a prospective, single-arm study to explore the efficacy and safety of SBRT Sequential CapeOX Regimen Chemotherapy Combined With Bevacizumab and Sintilimab in treatment with patients with initially unresectable advanced colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written Informed Consent Form (ICF) prior to any study specific procedures;
2. Age ≥ 18 years, ≤75 years;
3. Histologically or cytologically confirmed advanced Stage IV primary colorectal cancer,metastases cannot be removed;
4. No prior systemic treatment for advanced or metastatic colorectal cancer (including chemical therapy, epidermal growth factor receptor inhibitors such as cetuximab or panizumab, vascular endothelial growth factor inhibitors such as bevacizumab, immune checkpoint inhibitors such as anti-PD-1 or PD-L1 antibodies and anti-CTLA-4 antibodies);
5. The interval between adjuvant or neoadjuvant chemotherapy is more than one year;
6. According to the definition of RECIST 1.1, the investigator determined that the patient had at least one measurable disease;
7. At least one lesion is suitable for SBRT according to the evaluation of the researchers;
8. Patients with brain metastasis who are asymptomatic or stable after local treatment are allowed to be enrolled as long as they meet the following conditions:

1) Measurable lesions outside the central nervous system; 2) No central nervous system symptoms or no exacerbation of symptoms for at least 2 weeks; 3) no glucocorticoid treatment or discontinuation of glucocorticoid treatment within 7 days prior to administration of the first study drug;

9.ECOG 0-1;

10. Life expectancy >3 months;

11. LVEF ≥50%;

12.Adequate organ function, subject will meet the following laboratory criteria:

1. Absolute value of neutrophil (ANC) ≥1.5x109/L.
2. Platelet ≥90×109/L.
3. Hemoglobin≥ 9 g/dL.
4. Total bilirubin ≤1.5× upper normal value (ULN); Or total bilirubin & GT; ULN but direct bilirubin ≤ ULN;
5. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤2.5×ULN (ALT or AST ≤5×ULN in patients with liver metastasis);
6. Serum creatinine ≤1.5×ULN and creatinine clearance rate (calculated by Cockcroft-Gault formula) ≥60 mL /min;
7. Good coagulation function, defined as international standardized ratio (INR) or prothrombin time (PT) ≤1.5 ULN;
8. Normal thyroid function, defined as thyroid stimulating hormone (TSH) within the normal range. If the baseline TSH is outside the normal range, subjects with total T3 (or FT3) and FT4 within the normal range may be enrolled;
9. Urinary protein <2 +; If urine protein ≥2+, the 24-hour urine protein quantification must be ≤1g.

13.Women of childbearing age must be willing to use adequate contraception during study drug therapy.

Exclusion Criteria:

1. Prior treatment with anti-PD-L1, anti-PD-L2 drugs, or drugs that target another stimulating or co-inhibiting T-cell receptor (e.g., CTLA-4, OX-40, CD137);
2. Symptomatic or high-risk obstruction, bleeding, perforation, pneumonia (including noninfectious pneumonia with prior hormone therapy and pneumonia patients under treatment), etc;
3. Other malignant diseases other than colorectal cancer were diagnosed within 5 years prior to first administration (excluding radical basal cell carcinoma of the skin, squamous carcinoma of the skin, and/or radical resected carcinoma in situ);
4. Subject is currently participating in an interventional clinical study or has been treated with another study drug or study device in the 4 weeks prior to initial dosing;
5. An active autoimmune disease requiring systemic therapy (e.g., palliative drugs, glucocorticoids, or immunosuppressants) has occurred within 2 years prior to first dosing. Alternative therapies (e.g. thyroxine, insulin, or physiologic glucocorticoids for adrenal or pituitary dysfunction) are not considered systemic;
6. Subjects were receiving systemic glucocorticoid therapy (excluding nasal spray, inhalation, or other topical glucocorticoid) or any other form of immunosuppressive therapy within 7 days prior to study initial dosing;
7. Active hemoptysis (cough up at least 2.5ml or 1/2 teaspoon blood at a time) within 3 months prior to administration of the drug in the first study;
8. Imaging shows tumor invasion/invasion of large vessels or bleeding tendency as assessed by investigator or radiologist;
9. Had major surgery within 4 weeks prior to administration of the first study drug (except for surgery for biopsy purposes) or expected to have major surgery during the study period;
10. Severe unhealed wounds, ulcers or fractures;
11. Current or recent use of aspirin (within 10 days prior to receiving the first study dose) for 10 consecutive days (> 325 mg/ day) or other non-steroidal anti-inflammatory drugs known to inhibit platelet function; Current or recent (within 10 days prior to receiving the first study dose) treatment with a full-dose oral or parenteral anticoagulant or thrombolysis agent for 10 consecutive days;
12. Hereditary bleeding tendency or coagulopathy;
13. Digestive diseases such as active gastrointestinal ulcer, ulcerative colitis, intestinal obstruction, or other conditions that the investigator determines may cause gastrointestinal bleeding or perforation
14. Allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation is known;
15. Known allergy to oxaliplatin, capecitabine, sindilizumab or bevacizumab active ingredients or excipients;
16. Patients with multiple factors affecting oral medication (such as inability to swallow, post-gastrointestinal resection, chronic diarrhea and intestinal obstruction);
17. Has not fully recovered from toxicity and/or complications associated with any intervention prior to initiation of treatment (i.e., ≤ grade 1 or baseline, excluding fatigue or hair loss);
18. Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive);
19. Untreated active hepatitis B;
20. Active HCV-infected subjects (HCV antibody positive and HCV-RNA level above the detection limit);
21. Received live vaccine within 30 days prior to initial administration (cycle 1, day 1);

    Note: Acceptance of injectable inactivated virus vaccine against seasonal influenza is permitted within 30 days prior to first administration; Intranasally administered live attenuated flu vaccines are not allowed.
22. Pregnant or lactating women;
23. Grade II or above peripheral neuropathy according to NCI CTCAE standards;
24. Patients undergoing strong CYP3A4 inducers;
25. The presence of any serious or uncontrollable systemic disease;
26. Any medical history or disease evidence that may interfere with the study results, prevent the subjects from participating fully in the study, abnormal values of treatment or laboratory tests, or other conditions that the investigator considers inappropriate for the study because of other potential risks that the investigator considers inappropriate for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 12 months
  CR + PR rate according to the RECIST version 1.1 guidelines.
AEs | up to 36 months
  Adverse reactions refer to the occurrence and development of diseases in the process of using drugs according to normal usage and dosage to prevent, diagnose or treat diseases.Adverse reactions unrelated to the purpose of treatment.

SECONDARY OUTCOMES:
Disease control rate (DCR) | up to 12 months
  Disease control rate (DCR):CR + PR + SD rate according to the RECIST version 1.1 guidelines.
Progression-free survival (PFS) | up to 18 months
  To assess the efficacy of Tislelizumab Combined With Fruquintinib and SBRT for patients with advanced colorectal cancer by assessment of progression free survival (PFS) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Overall survival (OS) | up to 36 months
  The time interval between the start date of study drug and the date of death (any cause)

CONTACTS AND LOCATIONS:
Locations (1):
- Xianglin Yuan, Wuhan, Hubei, China